CLINICAL TRIAL: NCT01950819
Title: A 24 Month, Multicenter, Randomized, Open-label Safety and Efficacy Study of Concentration-controlled Everolimus With Reduced Calcineurin Inhibitor vs Mycophenolate With Standard Calcineurin Inhibitor in de Novo Renal Transplantation
Brief Title: Advancing Renal TRANSplant eFficacy and Safety Outcomes With an eveRolimus-based regiMen (TRANSFORM)
Acronym: TRANSFORM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001A2433; 2013-000322-66 (EudraCT Number); NCT02316938 (obsolete NCT alias)
Record Dates: First submitted 2013-08-20; First posted 2013-09-26 (Estimated); Results first posted 2019-01-30 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: End Stage Renal Disease (ESRD); Chronic Kidney Disease (CKD); Hemodialysis; Renal Replacement Therapy; Renal Transplantation
Keywords: kidney failure; dialysis; renal failure; transplantation
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic; Renal Insufficiency | interventions — Neoadjuvant Therapy; Basiliximab; thymoglobulin; Adrenal Cortex Hormones; Prednisone; Methylprednisolone; Everolimus; Cyclosporine; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Intervention Model Description: Open-label study
Oversight: Data Monitoring Committee: No

ARMS (2):
- EVR+rCNI (Experimental): Everolimus with reduced calcineurin inhibitor- everolimus (target trough level of 3-8 ng/mL) in combination with reduced exposure to CNI (cyclosporine or tacrolimus)
  Interventions: Biological: Induction therapy; Drug: Corticosteroids; Drug: EVR+rCNI
- MPA+sCNI (Active Comparator): Mycophenolate (mycophenolic acid sodium or mycophenolate mofetil) in combination with standard exposure to calcineurin inhibitor (cyclosporine or tacrolimus).
  Interventions: Biological: Induction therapy; Drug: Corticosteroids; Drug: MPA+sCNI

INTERVENTIONS:
Biological: Induction therapy — All subjects received induction therapy with basiliximab or rabbit anti-thymocyte globulin, in the peritransplant period.
  Other Names: Simulect, basiliximab, rATG, Thymoglobulin
Drug: Corticosteroids — All subjects received maintenance therapy with corticosteroids throughout the 24 month study period. A minimum dose of 5 mg prednisone, or equivalent, per day was maintained.
  Other Names: prednisone, methylprednisone, methylprednisolone, etc.
Drug: EVR+rCNI — Everolimus with reduced calcineurin inhibitor- everolimus (target trough level of 3-8 ng/mL) in combination with reduced exposure to CNI (cyclosporine or tacrolimus)
  Other Names: Zortress, Certican, Neoral, Prograf
  Arms: EVR+rCNI
Drug: MPA+sCNI — Mycophenolate (mycophenolic acid sodium or mycophenolate mofetil) in combination with standard exposure to calcineurin inhibitor (cyclosporine or tacrolimus).
  Other Names: Myfortic, Cellcept, Neoral, Prograf
  Arms: MPA+sCNI

SUMMARY:
This is a 2-year, randomized, multicenter, open-label, 2-arm study evaluating the graft function of everolimus and reduced CNI versus MPA and standard CNI in adult de novo renal transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained.
2. Subject randomized within 24 hr of completion of transplant surgery.
3. Recipient of a kidney with a cold ischemia time < 30 hours.
4. Recipient of a primary (or secondary, if first graft is not lost due to immunological reasons) renal transplant from a deceased heart beating, living unrelated, living related non-human leukocyte antigen identical or an expanded criteria donor.

Exclusion Criteria:

1. Subject unable to tolerate oral medication at time of randomization.
2. Use of other investigational drugs at the time of enrollment.
3. History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes.
4. Multi-organ transplant recipient.
5. Recipient of ABO incompatible allograft or complement-dependent lymphocytotoxic (CDC) crossmatch positive transplant.
6. Subject at high immunological risk for rejection as determined by local practice for assessment of anti-donor reactivity e.g. high PRA, presence of pre-existing DSA.
7. Subject who is HIV-positive.
8. HBsAg and/or a HCV positive subject with evidence of elevated LFTs (ALT/AST levels ≥ 2.5 times ULN). Viral serology results obtained within 6 months prior to randomization are acceptable.
9. Recipient of a kidney from a donor who tests positive for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or anti-hepatitis C virus (HCV).
10. Subject with a BMI greater than 35.
11. Subject with severe systemic infections, current or within the two weeks prior to randomization.
12. Subject requiring systemic anticoagulation.
13. History of malignancy of any organ system.
14. Subject with severe restrictive or obstructive pulmonary disorders.
15. Subject with severe hypercholesterolemia or hypertriglyceridemia that cannot be controlled.
16. Subject with white blood cell (WBC) count ≤ 2,000 /mm3 or with platelet count ≤ 50,000 /mm3.
17. Pregnant or nursing (lactating) women.
18. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using effective methods of contraception during dosing of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2037 (Actual)
Dates: Start 2013-12-03 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2018-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (165):
- United States (35):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Loma Linda, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Aurora, Colorado
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Burlington, Massachusetts
  - Novartis Investigative Site, Ann Arbor, Michigan
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Livingston, New Jersey
  - Novartis Investigative Site, Buffalo, New York
  - Novartis Investigative Site, The Bronx, New York
  - Novartis Investigative Site, Chapel Hill, North Carolina
  - Novartis Investigative Site, Durham, North Carolina
  - Novartis Investigative Site, Winston-Salem, North Carolina
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Harrisburg, Pennsylvania
  - Novartis Investigative Site, Providence, Rhode Island
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Fort Worth, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Salt Lake City, Utah
  - Novartis Investigative Site, Charlottesville, Virginia
  - Novartis Investigative Site, Seattle, Washington
  - Novartis Investigative Site, Madison, Wisconsin
  - Novartis Investigative Site, Milwaukee, Wisconsin
- Argentina (6):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, San Martín, Buenos Aires
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Corrientes
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Santa Fe
- Australia (10):
  - Novartis Investigative Site, Camperdown, New South Wales
  - Novartis Investigative Site, Randwick, New South Wales
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, Woolloongabba, Queensland
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Clayton, Victoria
  - Novartis Investigative Site, Heidelberg, Victoria
  - Novartis Investigative Site, Parkville, Victoria
  - Novartis Investigative Site, Murdoch, Western Australia
  - Novartis Investigative Site, Nedlands, Western Australia
- Austria (2):
  - Novartis Investigative Site, Innsbruck, Tyrol
  - Novartis Investigative Site, Linz
- Belgium (4):
  - Novartis Investigative Site, Edegem, Antwerpen
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
- Brazil (2):
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, São Paulo, São Paulo
- Novartis Investigative Site, Sofia, BGR, Bulgaria
- Novartis Investigative Site, Santiago, Chile
- Colombia (2):
  - Novartis Investigative Site, Cali, Valle del Cauca Department
  - Novartis Investigative Site, Bogotá
- Croatia (2):
  - Novartis Investigative Site, Rijeka
  - Novartis Investigative Site, Zagreb
- Czechia (2):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Prague
- Novartis Investigative Site, Al Mansurah, Egypt
- France (5):
  - Novartis Investigative Site, Nice, Cedex1
  - Novartis Investigative Site, Tours, Indre Et Loire
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Reims
- Germany (10):
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Hannover Muenden
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Kaiserslautern
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, München
- Greece (3):
  - Novartis Investigative Site, Thessaloniki, GR
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Pátrai
- India (4):
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Vellore, Tamil Nadu
- Israel (2):
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Tel Aviv
- Italy (9):
  - Novartis Investigative Site, Bari, BA
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Parma, PR
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Novara
- Japan (3):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Toyoake, Aichi-ken
  - Novartis Investigative Site, Chiba, Chiba
- Novartis Investigative Site, Kuwait City, Kuwait
- Lebanon (2):
  - Novartis Investigative Site, El Achrafiyé
  - Novartis Investigative Site, Saida
- Malaysia (2):
  - Novartis Investigative Site, Kuala Lumpur
  - Novartis Investigative Site, Selangor Darul Ehsan
- Novartis Investigative Site, Guadalajara, Jalisco, Mexico
- Netherlands (6):
  - Novartis Investigative Site, Maastricht, AZ
  - Novartis Investigative Site, Utrecht, The Netherlands
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Leiden
  - Novartis Investigative Site, Nijmegen
- Novartis Investigative Site, Oslo, Norway
- Novartis Investigative Site, Quezon City, Philippines
- Poland (3):
  - Novartis Investigative Site, Szczecin, Pomeranian Voivodeship
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Poznan
- Portugal (4):
  - Novartis Investigative Site, Carnaxide, Lisbon District
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Porto
- Russia (5):
  - Novartis Investigative Site, Krasnodar
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Volzhskiy
  - Novartis Investigative Site, Yekaterinburg
- Saudi Arabia (3):
  - Novartis Investigative Site, Dammam
  - Novartis Investigative Site, Jeddah
  - Novartis Investigative Site, Riyadh
- Serbia (3):
  - Novartis Investigative Site, Belgrade
  - Novartis Investigative Site, Niš
  - Novartis Investigative Site, Novi Sad
- Novartis Investigative Site, Singapore, Singapore
- Slovakia (4):
  - Novartis Investigative Site, Banská Bystrica
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Martin
- Novartis Investigative Site, Ljubljana, Slovenia
- Novartis Investigative Site, Cape Town, Western Province, South Africa
- South Korea (2):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Spain (8):
  - Novartis Investigative Site, Granada, Andalusia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Zaragoza
- Sweden (3):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Uppsala
- Novartis Investigative Site, Bern, Switzerland
- Taiwan (3):
  - Novartis Investigative Site, Tainan, Taiwan ROC
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
- Thailand (2):
  - Novartis Investigative Site, Ratchathewi, Bangkok
  - Novartis Investigative Site, Bangkok
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Antalya
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Mecidiyekoy/Istanbul

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydata request.com

REFERENCES:
- [Derived] Aubert O, Divard G, Pascual J, Oppenheimer F, Sommerer C, Citterio F, Tedesco H, Chadban S, Henry M, Vincenti F, Srinivas T, Watarai Y, Legendre C, Bernhardt P, Loupy A. Application of the iBox prognostication system as a surrogate endpoint in the TRANSFORM randomised controlled trial: proof-of-concept study. BMJ Open. 2021 Oct 7;11(10):e052138. doi: 10.1136/bmjopen-2021-052138. PMID 34620664
- [Derived] Watarai Y, Danguilan R, Casasola C, Chang SS, Ruangkanchanasetr P, Kee T, Wong HS, Kenmochi T, Amante AJ, Shu KH, Ingsathit A, Bernhardt P, Hernandez-Gutierrez MP, Han DJ, Kim MS. Everolimus-facilitated calcineurin inhibitor reduction in Asian de novo kidney transplant recipients: 2-year results from the subgroup analysis of the TRANSFORM study. Clin Transplant. 2021 Oct;35(10):e14415. doi: 10.1111/ctr.14415. Epub 2021 Sep 23. PMID 34216395
- [Derived] Citterio F, Henry M, Kim DY, Kim MS, Han DJ, Kenmochi T, Mor E, Tisone G, Bernhardt P, Hernandez Gutierrez MP, Watarai Y. Wound healing adverse events in kidney transplant recipients receiving everolimus with reduced calcineurin inhibitor exposure or current standard-of-care: insights from the 24-month TRANSFORM study. Expert Opin Drug Saf. 2020 Oct;19(10):1339-1348. doi: 10.1080/14740338.2020.1792441. Epub 2020 Jul 20. PMID 32633157
- [Derived] Berger SP, Sommerer C, Witzke O, Tedesco H, Chadban S, Mulgaonkar S, Qazi Y, de Fijter JW, Oppenheimer F, Cruzado JM, Watarai Y, Massari P, Legendre C, Citterio F, Henry M, Srinivas TR, Vincenti F, Gutierrez MPH, Marti AM, Bernhardt P, Pascual J; TRANSFORM investigators. Two-year outcomes in de novo renal transplant recipients receiving everolimus-facilitated calcineurin inhibitor reduction regimen from the TRANSFORM study. Am J Transplant. 2019 Nov;19(11):3018-3034. doi: 10.1111/ajt.15480. Epub 2019 Jul 1. PMID 31152476
- [Derived] Pascual J, Berger SP, Witzke O, Tedesco H, Mulgaonkar S, Qazi Y, Chadban S, Oppenheimer F, Sommerer C, Oberbauer R, Watarai Y, Legendre C, Citterio F, Henry M, Srinivas TR, Luo WL, Marti A, Bernhardt P, Vincenti F; TRANSFORM Investigators. Everolimus with Reduced Calcineurin Inhibitor Exposure in Renal Transplantation. J Am Soc Nephrol. 2018 Jul;29(7):1979-1991. doi: 10.1681/ASN.2018010009. Epub 2018 May 11. PMID 29752413

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The full analysis set consisted of all randomized and transplanted patients. The safet set consisted of all patients who received at least one dose of study drug
Pre-assignment Details: 2226 patients screened; 2037 patients transplanted and randomized to treatment.
Period: Overall Study
Arm/Group | EVR+rCNI | MPA+sCNI
Started | 1022 | 1015
Completed | 893 | 881
Not Completed | 129 | 134
Not completed — Graft Loss | 35 | 30
Not completed — Death | 29 | 34
Not completed — Subject / Gardian decision | 54 | 51
Not completed — technical problems | 2 | 0
Not completed — Pregnancy | 0 | 2
Not completed — Lost to Follow-up | 9 | 17

BASELINE CHARACTERISTICS:
Population: Full Analysis set
Groups:
- Total: Total of all reporting groups
Arm/Group | EVR+rCNI | MPA+sCNI | Total
Number analyzed (Participants) | 1022 | 1015 | 2037
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: full analysis set
  years | 48.79 (14.123) | 48.75 (14.515) | 48.77 (14.316)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: full analysis set
  Participants
    Female | 312 | 308 | 620
    Male | 710 | 707 | 1417
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity Population: full analysis set
  Participants
    Hispany or Latino | 157 | 132 | 289
    not Hispanic or Latino | 646 | 661 | 1307
    Unknown or not reported | 219 | 222 | 441
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race Population: full analysis set
  Participants
    Caucasian | 743 | 735 | 1478
    Asian | 136 | 157 | 293
    Black | 43 | 35 | 78
    Other | 100 | 88 | 188

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Failure on the Composite of Treated Biopsy-proven Acute Rejection (tBPAR) or Estimated Glomerular Filtration Rate (eGFR) < 50 mL/Min/1.73m2.
Description: Incidence of failure on the composite of treated biopsy-proven acute rejection (tBPAR) or estimated glomerular filtration rate (eGFR) < 50 mL/min/1.73m2.
Time Frame: Month 12 is Primary, Month 24 secondary
Population: full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | EVR+rCNI | MPA+sCNI
Number analyzed (Participants) | 1022 | 1015
Participants
  month 12 | 489 | 456
  month 24 | 489 | 443
Statistical Analysis 1: Comparison: EVR+rCNI vs MPA+sCNI; calculated at month 12; Test type: Non-Inferiority — p vale for non inferiority margin is 10 %; p = 0.001, Logistic Regression Model; Odds Ratio (OR) = 3.0, 95% CI 2-sided [-1.4 to 7.3]

2. Secondary Outcome: Incidence of Failure on the Composite of (Treated Biopsy Proven Acute Rejection (tBPAR), Graft Loss or Death
Description: Incidence of failure on the composite of (treated biopsy proven acute rejection (tBPAR), graft loss or death
Time Frame: Month 12 and 24
Population: full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | EVR+rCNI | MPA+sCNI
Number analyzed (Participants) | 1022 | 1015
Participants
  month 12 | 146 | 131
  month 24 | 169 | 147

3. Secondary Outcome: Incidence of Failure on the Composite Endpoint of tBPAR, Graft Loss, Death or eGFR < 50 mL/Min/1.73m2
Description: Incidence of failure on the composite endpoint of tBPAR, graft loss, death or eGFR < 50 mL/min/1.73m2
Time Frame: Month 12 and 24
Population: full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | EVR+rCNI | MPA+sCNI
Number analyzed (Participants) | 1022 | 1015
Participants
  month 12 | 497 | 466
  month 24 | 497 | 457

4. Secondary Outcome: Incidence of Failure on the Composite Endpoint of Graft Loss or Death.
Description: Incidence of failure on the composite endpoint of graft loss or death.
Time Frame: Month 12 and 24
Population: full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | EVR+rCNI | MPA+sCNI
Number analyzed (Participants) | 1022 | 1015
Participants
  month 12 | 51 | 54
  month 24 | 67 | 65

5. Secondary Outcome: Incidence of Death, Graft Loss, tBPAR, BPAR, tAR, AR and Humoral Rejection
Description: Incidence of death, graft loss, tBPAR (treated biopsy proven acute rejection), BPAR (biopsy proven acute rejection), tAR (treated acute rejection), AR (acute rejection) and humoral rejection (aAMR : active antibody mediated rejection and cAMR: chronic antibody mediated rejection)
Time Frame: Month 12 and 24
Population: full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | EVR+rCNI | MPA+sCNI
Number analyzed (Participants) | 1022 | 1015
Participants
  deaths month 12 | 20 | 28
  deaths month 24 | 32 | 36
  graft loss month 12 | 33 | 28
  graft loss month 24 | 37 | 32
  tBPAR month 12 | 107 | 91
  tBPAR month 24 | 118 | 98
  BPAR month 12 | 114 | 95
  BPAR month 24 | 127 | 104
  tAR month 12 | 129 | 117
  tAR month 24 | 145 | 126
  AR month 12 | 147 | 133
  AR month 24 | 167 | 144
  aAMR month 12 | 73 | 61
  aAMR month 24 | 84 | 69
  cAMR month 12 | 9 | 14
  cAMR month 24 | 13 | 18

6. Secondary Outcome: Incidence of eGFR < 50 mL/Min/1.73m2
Description: Incidence of eGFR < 50 mL/min/1.73m2
Time Frame: Month 12 and 24
Population: full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | EVR+rCNI | MPA+sCNI
Number analyzed (Participants) | 1022 | 1015
Participants
  month 12 | 456 | 424
  month 24 | 474 | 423

7. Secondary Outcome: Renal Allograft Function : Mean Estimated Glomerular Filtration Rate, eGFR
Description: Renal allograft function : mean estimated glomerular filtration rate, eGFR
Time Frame: Baseline (week 4), Month 12 and 24
Population: full analysis set
Measure: Mean (Standard Error); unit: mL/min/1.73m2
Arm/Group | EVR+rCNI | MPA+sCNI
Number analyzed (Participants) | 1022 | 1015
mL/min/1.73m2
  baseline (week 4) | 53.13 (0.765) | 52.25 (0.684)
  month 12 | 53.29 (0.698) | 54.49 (0.667)
  month 24 | 52.63 (0.744) | 54.91 (0.719)

8. Secondary Outcome: Evolution of Renal Function, as eGFR, Over Time by Slope Analysis.
Description: Rate of change of renal function, as eGFR, calculated using MDRD4 formula (Coresh, 2003) and adjusted by covariates.
Time Frame: Month 12 and 24
Population: full analysis set
Measure: Mean (Standard Error); unit: mL / min / 1.73m2 / day
Arm/Group | EVR+rCNI | MPA+sCNI
Number analyzed (Participants) | 1022 | 1015
mL / min / 1.73m2 / day | 0.0001 (0.0008) | 0.0047 (0.0008)

9. Secondary Outcome: Renal Function Assessed by Creatinine Lab Values
Description: Mean Renal function as assessed in clinical practice, by ceatinine values. Analysis is done without considering missing values for analysis.
Time Frame: Month 12 and 24
Population: full analysis set with measure
Measure: Mean (Standard Deviation); unit: micromol/L
Arm/Group | EVR+rCNI | MPA+sCNI
Number analyzed (Participants) | 1022 | 1015
micromol/L
  screening baseline (creatinine, micromol/L): number analyzed (Participants) | 448 | 498
  screening baseline (creatinine, micromol/L) | 590.1 (262.78) | 601.8 (265.08)
  month 12 (creatinine, micromol/L): number analyzed (Participants) | 742 | 816
  month 12 (creatinine, micromol/L) | 129.8 (49.12) | 128.6 (50.80)
  month 24 (creatinine, micromol/L): number analyzed (Participants) | 640 | 719
  month 24 (creatinine, micromol/L) | 130.1 (53.54) | 127.6 (52.50)

10. Secondary Outcome: Renal Function by Alternative Formulae (e.g. CKD-EPI). eGFR Values Reported
Description: Mean Renal function as used in clinical practice, using different formula for calculation of renal function than MDRD4 (our primary efficacy parameter), and other alternate formulae (e.g. CKD-EPI). Analysis is done without considering missing values for analysis.
Time Frame: Month 12 and 24
Population: full analysis set with measure
Measure: Mean (Standard Deviation); unit: mL/min/1.73m2
Arm/Group | EVR+rCNI | MPA+sCNI
Number analyzed (Participants) | 1022 | 1015
mL/min/1.73m2
  eGFR (Hoek) baseline (mL/min/1.73m2): number analyzed (Participants) | 443 | 493
  eGFR (Hoek) baseline (mL/min/1.73m2) | 21.38 (14.296) | 20.10 (12.408)
  eGFR (Hoek) month 12 (mL/min/1.73m2): number analyzed (Participants) | 734 | 801
  eGFR (Hoek) month 12 (mL/min/1.73m2) | 50.08 (14.430) | 52.00 (14.533)
  eGFR (Hoek) month 24 (mL/min/1.73m2): number analyzed (Participants) | 641 | 702
  eGFR (Hoek) month 24 (mL/min/1.73m2) | 49.86 (14.604) | 52.75 (15.406)
  eGFR (MDRD4) baseline (mL/min/1.73m2): number analyzed (Participants) | 448 | 498
  eGFR (MDRD4) baseline (mL/min/1.73m2) | 11.79 (8.697) | 11.56 (8.853)
  eGFR (MDRD4) month 12 (mL/min/1.73m2): number analyzed (Participants) | 742 | 816
  eGFR (MDRD4) month 12 (mL/min/1.73m2) | 57.59 (19.685) | 57.58 (18.768)
  eGFR (MDRD4) month 24 (mL/min/1.73m2): number analyzed (Participants) | 640 | 719
  eGFR (MDRD4) month 24 (mL/min/1.73m2) | 58.07 (20.168) | 58.68 (19.541)
  eGFR-CKDEPI baseline (mL/min/1.73m2): number analyzed (Participants) | 448 | 498
  eGFR-CKDEPI baseline (mL/min/1.73m2) | 11.29 (9.094) | 11.05 (9.195)
  eGFR-CKDEPI month 12(mL/min/1.73m2): number analyzed (Participants) | 742 | 816
  eGFR-CKDEPI month 12(mL/min/1.73m2) | 58.83 (20.686) | 58.75 (19.757)
  eGFR-CKDEPI month 24 (mL/min/1.73m2): number analyzed (Participants) | 640 | 719
  eGFR-CKDEPI month 24 (mL/min/1.73m2) | 59.39 (21.077) | 59.95 (20.652)

11. Secondary Outcome: Incidence of Adverse Events, Serious Adverse Events and Adverse Events Leading to Study Regimen Discontinuation.
Description: Incidence of adverse events, serious adverse events and adverse events leading to study regimen discontinuation.
Time Frame: Month 24
Population: safety set 24 months analysis
Measure: Count of Participants; unit: Participants
Arm/Group | EVR+rCNI | MPA+sCNI
Number analyzed (Participants) | 1014 | 1012
Participants | 276 | 152

12. Secondary Outcome: Incidence of Cytomegalovirus and BK Virus, New Onset Diabetes Mellitus, Chronic Kidney Disease With Associated Proteinuria and Calcineurin Inhibitor Associated Adverse Events.
Description: Incidence of cytomegalovirus and BK virus, new onset diabetes mellitus, chronic kidney disease with associated proteinuria and calcineurin inhibitor associated adverse events.
Time Frame: Month 24
Population: safety set
Measure: Count of Participants; unit: Participants
Arm/Group | EVR+rCNI | MPA+sCNI
Number analyzed (Participants) | 1014 | 1012
Participants
  clinical signs of CMV infection | 53 | 132
  any BKV infection | 103 | 154
  new onset of diabetes mellitus | 144 | 138
  at least one event of interest | 871 | 764

13. Secondary Outcome: Urinary Protein and Albumin Excretion by Treatment Estimated by Urinary Protein/Creatinine and Urinary Albumin/Creatinine Ratios.
Description: Mean urinary protein and albumin excretion by treatment estimated by mean urinary protein/creatinine and urinary albumin/creatinine ratios.
Time Frame: Baseline, Month 12 and 24
Population: safety set with measure
Measure: Mean (Standard Deviation); unit: mg/g
Arm/Group | EVR+rCNI | MPA+sCNI
Number analyzed (Participants) | 1014 | 1012
mg/g
  albumine /creatinine ratio baseline: number analyzed (Participants) | 79 | 54
  albumine /creatinine ratio baseline | 1019.75 (2737.96) | 646.111 (799.234)
  albumine /creatinine ratio month 12: number analyzed (Participants) | 729 | 794
  albumine /creatinine ratio month 12 | 150.061 (482.394) | 111.322 (444.631)
  albumine /creatinine ratio month 24: number analyzed (Participants) | 633 | 708
  albumine /creatinine ratio month 24 | 149.049 (464.470) | 116.618 (433.392)
  protein /creatinine ratio baseline: number analyzed (Participants) | 79 | 54
  protein /creatinine ratio baseline | 1648.10 (3768.22) | 1142.59 (1003.69)
  protein /creatinine ratio month 12: number analyzed (Participants) | 729 | 794
  protein /creatinine ratio month 12 | 298.557 (642.103) | 234.698 (583.632)
  protein /creatinine ratio month 24: number analyzed (Participants) | 633 | 708
  protein /creatinine ratio month 24 | 290.242 (588.119) | 233.009 (524.383)

14. Secondary Outcome: Incidence of Major Cardiovascular Events.
Description: Incidence of major cardiovascular events by Preferred Term
Time Frame: Month 24
Population: safety set
Measure: Count of Participants; unit: Participants
Arm/Group | EVR+rCNI | MPA+sCNI
Number analyzed (Participants) | 1014 | 1012
Participants | 66 | 86

15. Secondary Outcome: Incidence of Malignancies.
Description: Incidence of malignancies.
Time Frame: Month 24
Population: safety set
Measure: Count of Participants; unit: Participants
Arm/Group | EVR+rCNI | MPA+sCNI
Number analyzed (Participants) | 1014 | 1012
Participants | 41 | 39

16. Secondary Outcome: Incidence of Failure on the Composite of Treated Biopsy-proven Acute Rejection (tBPAR) or Estimated Glomerular Filtration Rate (eGFR) < 50 mL/Min/1.73m2 Among Compliant Subjects.
Description: Incidence of failure on the composite of treated biopsy-proven acute rejection (tBPAR) or estimated glomerular filtration rate (eGFR) < 50 mL/min/1.73m2 among compliant subjects.
Time Frame: Month 12 and 24
Population: compliance set
Measure: Count of Participants; unit: Participants
Arm/Group | EVR+rCNI | MPA+sCNI
Number analyzed (Participants) | 187 | 277
Participants
  month 12 | 60 | 106
  month 24 | 62 | 102

17. Secondary Outcome: Incidence tBPAR (Treated Biopsy-proven Acute Rejection) by Severity and Time to Event (Participants)
Description: Incidence tBPAR, defined as any condition where the subject received anti-rejection treatment and was histologically diagnosed as acute rejection (according to the Banff 2009 criteria), by severity (grade IA, IB, IIA, IIB, III) and time to event. Grades for T-cell mediated rejection, with increasing severity:
  * Type IA - Significant interstitial infiltration (> 25% of parenchyma) and foci of moderate tubulitis (> 4 mononuclear cells/tubular cross section or group of 10 tubular cells).
  * Type IB - Significant interstitial infiltration (> 25% of parenchyma) and foci of severe tubulitis (> 10 mononuclear cells/tubular cross section or group of 10 tubular cells).
  * Type IIA - Mild to moderate intimal arteritis
  * Type IIB - Severe intimal arteritis comprising > 25% of the lumenal area
  * Type III - Transmural (full vessel wall thickness) arteritis and/or arterial fibrinoid change and necrosis of medial smooth muscle cells (with accompanying lymphocytic inflammation)
Time Frame: Month 12 and 24
Population: full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | EVR+rCNI | MPA+sCNI
Number analyzed (Participants) | 1022 | 1015
Participants
  Patient's maximum tBPAR grade : no grade (missing) | 25 | 18
  Patient's maximum tBPAR grade : grade IA | 34 | 36
  Patient's maximum tBPAR grade : grade IB | 23 | 17
  Patient's maximum tBPAR grade : grade IIA | 21 | 24
  Patient's maximum tBPAR grade : grade IIB | 9 | 3
  Patient's maximum tBPAR grade : grade III | 6 | 0

18. Secondary Outcome: Incidence tBPAR (Treated Biopsy-proven Acute Rejection) by Severity and Time to Event (Events)
Description: as for outcome 17
Time Frame: Month 12 and 24
Population: full analysis set
Measure: Number; unit: events
Arm/Group | EVR+rCNI | MPA+sCNI
Number analyzed (Participants) | 1022 | 1015
events
  overall number of tBPAR regardless of grade | 146 | 116
  number of tBPAR regardless of grade days 1-90 | 72 | 63
  number of tBPAR regardless of grade days 91-180 | 24 | 14
  number of tBPAR regardless of grade days 181-360 | 25 | 20
  number of tBPAR regardless of grade days 361-540 | 12 | 15
  number of tBPAR regardless of grade days 541-720 | 11 | 2
  number of tBPAR regardless of grade days 721-810 | 2 | 2

19. Secondary Outcome: Incidence of tBPAR (Treated Biopsy-proven Acute Rejection) Excluding Grade IA Rejections
Description: Incidence of tBPAR, defined as any condition where the subject received anti-rejection treatment and was histologically diagnosed as acute rejection (according to the Banff 2009 criteria), excluding grade IA rejections. Grades for T-cell mediated rejection, with increasing severity:
  * Type IA - Significant interstitial infiltration (> 25% of parenchyma) and foci of moderate tubulitis (> 4 mononuclear cells/tubular cross section or group of 10 tubular cells).
  * Type IB - Significant interstitial infiltration (> 25% of parenchyma) and foci of severe tubulitis (> 10 mononuclear cells/tubular cross section or group of 10 tubular cells).
  * Type IIA - Mild to moderate intimal arteritis
  * Type IIB - Severe intimal arteritis comprising > 25% of the lumenal area
  * Type III - Transmural (full vessel wall thickness) arteritis and/or arterial fibrinoid change and necrosis of medial smooth muscle cells (with accompanying lymphocytic inflammation)
Time Frame: Month 12 and 24
Population: full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | EVR+rCNI | MPA+sCNI
Number analyzed (Participants) | 1022 | 1015
Participants
  month 12 | 66 | 53
  month 24 | 74 | 55

20. Secondary Outcome: Incidence of Composite of tBPAR (Treated Biopsy-proven Acute Rejection)or eGRF<50 mL/Min/1.73m2 by Subgroup
Description: Incidence of composite of tBPAR or eGRF<50 mL/min/1.73m2 by subgroup
Time Frame: Month 12 and 24
Population: full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | EVR+rCNI | MPA+sCNI
Number analyzed (Participants) | 1022 | 1015
Participants
  month 12 | 489 | 456
  month 24 | 489 | 443

21. Secondary Outcome: Incidence of tBPAR (Excluding Grade IA Rejections) or GFR<50 mL/Min/1.73m2
Description: Incidence of tBPAR (excluding grade IA rejections) or GFR<50 mL/min/1.73m2
Time Frame: Month 12 and 24
Population: full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | EVR+rCNI | MPA+sCNI
Number analyzed (Participants) | 1022 | 1015
Participants
  month 12 | 475 | 441
  month 24 | 475 | 426

22. Secondary Outcome: Incidence of Failure on the Composite of (Treated Biopsy Proven Acute Rejection (tBPAR), Graft Loss or Death or Loss to Follow-up
Description: Incidence of failure on the composite of (treated biopsy proven acute rejection (tBPAR), graft loss or death or loss to follow-up
Time Frame: Month 12 and 24
Population: full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | EVR+rCNI | MPA+sCNI
Number analyzed (Participants) | 1022 | 1015
Participants
  month 12 | 181 | 170
  month 24 | 218 | 201

ADVERSE EVENTS:
Time Frame: Adverse Events are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All Adverse events are reported in this record from First Patient First Treatment until Last Patient Last Visit up to approximately 4 years.
Description: treatment emergent AE / SAE . Consistent with EudraCT disclosure specifications, Novartis has reported under the Serious adverse events fields "number of deaths resulting from adverse events" all those deaths, resulting from serious adverse events that are deemed to be causally related to treatment by the investigator.
Groups:
- Everolimus Plus@Reduced CNI: Everolimus plus@reduced CNI
- MPA Plus Standard@CNI: MPA plus standard@CNI
Arm/Group | Everolimus Plus@Reduced CNI | MPA Plus Standard@CNI
All-Cause Mortality (participants affected / at risk) | 20/1014 | 29/1012
Serious Adverse Events (participants affected / at risk) | 593/1014 | 613/1012
Other Adverse Events (participants affected / at risk) | 951/1014 | 942/1012
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus Plus@Reduced CNI (N=1014) | MPA Plus Standard@CNI (N=1012)
Agranulocytosis (Blood and lymphatic system disorders) | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 14 | 6
Atypical haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 1 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 5
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 1
Haemolysis (Blood and lymphatic system disorders) | 2 | 0
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 1 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 4 | 12
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Lymphatic obstruction (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 6
Pancytopenia (Blood and lymphatic system disorders) | 2 | 1
Polycythaemia (Blood and lymphatic system disorders) | 0 | 2
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 1 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 1
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 8 | 3
Acute coronary syndrome (Cardiac disorders) | 4 | 2
Acute myocardial infarction (Cardiac disorders) | 6 | 6
Angina pectoris (Cardiac disorders) | 6 | 5
Angina unstable (Cardiac disorders) | 1 | 1
Aortic valve stenosis (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 12 | 12
Atrial flutter (Cardiac disorders) | 4 | 1
Bradycardia (Cardiac disorders) | 3 | 1
Cardiac arrest (Cardiac disorders) | 4 | 4
Cardiac asthma (Cardiac disorders) | 0 | 1
Cardiac dysfunction (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 9 | 7
Cardiac failure acute (Cardiac disorders) | 2 | 0
Cardiac failure chronic (Cardiac disorders) | 2 | 1
Cardiac failure congestive (Cardiac disorders) | 6 | 3
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Cardiorenal syndrome (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 2 | 6
Coronary artery insufficiency (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 2 | 1
Hypertensive heart disease (Cardiac disorders) | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 1 | 0
Left ventricular hypertrophy (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 5 | 6
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0
Pericarditis constrictive (Cardiac disorders) | 0 | 1
Pulseless electrical activity (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 2
Ventricular extrasystoles (Cardiac disorders) | 0 | 1
Ventricular tachyarrhythmia (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 1
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 | 1
Congenital megaureter (Congenital, familial and genetic disorders) | 1 | 0
Hydrocele (Congenital, familial and genetic disorders) | 1 | 2
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 0 | 1
Mastoid effusion (Ear and labyrinth disorders) | 1 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Goitre (Endocrine disorders) | 1 | 0
Hyperparathyroidism (Endocrine disorders) | 1 | 0
Hyperparathyroidism tertiary (Endocrine disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 3
Glaucoma (Eye disorders) | 0 | 1
Optic ischaemic neuropathy (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 4 | 2
Abdominal pain (Gastrointestinal disorders) | 9 | 14
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 4 | 3
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 1
Acute abdomen (Gastrointestinal disorders) | 1 | 0
Anal polyp (Gastrointestinal disorders) | 1 | 0
Anogenital dysplasia (Gastrointestinal disorders) | 0 | 1
Barrett's oesophagus (Gastrointestinal disorders) | 1 | 0
Chronic gastritis (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 3
Crohn's disease (Gastrointestinal disorders) | 1 | 1
Diabetic gastroparesis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 27 | 55
Diverticulum (Gastrointestinal disorders) | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 2
Duodenal perforation (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Encapsulating peritoneal sclerosis (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 2 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Gastrointestinal fistula (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Hernial eventration (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 5 | 2
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 2 | 5
Intestinal obstruction (Gastrointestinal disorders) | 2 | 2
Intestinal perforation (Gastrointestinal disorders) | 2 | 1
Intra-abdominal fluid collection (Gastrointestinal disorders) | 5 | 1
Intra-abdominal haematoma (Gastrointestinal disorders) | 2 | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Lumbar hernia (Gastrointestinal disorders) | 0 | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 3 | 9
Oesophageal achalasia (Gastrointestinal disorders) | 1 | 0
Oesophageal spasm (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 2
Pancreatitis acute (Gastrointestinal disorders) | 0 | 2
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2
Retching (Gastrointestinal disorders) | 0 | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 2 | 5
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 1
Salivary gland enlargement (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 4
Stomatitis (Gastrointestinal disorders) | 0 | 2
Umbilical hernia (Gastrointestinal disorders) | 3 | 0
Volvulus (Gastrointestinal disorders) | 1 | 0
Volvulus of small bowel (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 6 | 13
Asthenia (General disorders) | 0 | 1
Catheter site haemorrhage (General disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 2
Chills (General disorders) | 1 | 2
Death (General disorders) | 0 | 2
Fatigue (General disorders) | 2 | 2
Gait inability (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 0 | 1
Generalised oedema (General disorders) | 1 | 0
Hyperthermia (General disorders) | 1 | 0
Hypothermia (General disorders) | 0 | 1
Ill-defined disorder (General disorders) | 0 | 1
Impaired healing (General disorders) | 10 | 1
Malaise (General disorders) | 2 | 1
Medical device site discomfort (General disorders) | 1 | 0
Medical device site inflammation (General disorders) | 1 | 0
Microlithiasis (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 2
Oedema peripheral (General disorders) | 7 | 4
Pain (General disorders) | 0 | 1
Peripheral swelling (General disorders) | 0 | 2
Pyrexia (General disorders) | 35 | 36
Sudden death (General disorders) | 1 | 0
Suprapubic pain (General disorders) | 0 | 1
Swelling (General disorders) | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 1 | 2
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 1
Biliary dilatation (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 3
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 2
Cholestasis (Hepatobiliary disorders) | 1 | 0
Hepatocellular injury (Hepatobiliary disorders) | 0 | 1
Perforation bile duct (Hepatobiliary disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1
Chronic allograft nephropathy (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Immunosuppression (Immune system disorders) | 1 | 0
Kidney transplant rejection (Immune system disorders) | 18 | 17
Renal transplant failure (Immune system disorders) | 4 | 5
Transplant rejection (Immune system disorders) | 45 | 25
Abdominal abscess (Infections and infestations) | 1 | 1
Abdominal infection (Infections and infestations) | 1 | 0
Actinomycosis (Infections and infestations) | 1 | 0
Adenoviral haemorrhagic cystitis (Infections and infestations) | 0 | 1
Adenovirus infection (Infections and infestations) | 2 | 1
Anal abscess (Infections and infestations) | 1 | 1
Appendicitis (Infections and infestations) | 0 | 3
Arteriovenous fistula site infection (Infections and infestations) | 0 | 1
Arthritis bacterial (Infections and infestations) | 0 | 1
Arthritis infective (Infections and infestations) | 1 | 0
Asymptomatic bacteriuria (Infections and infestations) | 1 | 0
Atypical pneumonia (Infections and infestations) | 2 | 0
BK virus infection (Infections and infestations) | 3 | 5
Bacteraemia (Infections and infestations) | 3 | 0
Bacterial diarrhoea (Infections and infestations) | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 1
Bacterial prostatitis (Infections and infestations) | 1 | 1
Bacterial pyelonephritis (Infections and infestations) | 2 | 1
Bacterial sepsis (Infections and infestations) | 1 | 1
Bacteriuria (Infections and infestations) | 0 | 2
Blister infected (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 3
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 2
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0
Candida infection (Infections and infestations) | 2 | 0
Candiduria (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 5 | 6
Chest wall abscess (Infections and infestations) | 0 | 1
Chronic sinusitis (Infections and infestations) | 1 | 0
Chronic tonsillitis (Infections and infestations) | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 4 | 3
Clostridium difficile infection (Infections and infestations) | 1 | 0
Corona virus infection (Infections and infestations) | 1 | 0
Cryptococcosis (Infections and infestations) | 0 | 3
Cystitis viral (Infections and infestations) | 1 | 0
Cytomegalovirus colitis (Infections and infestations) | 0 | 9
Cytomegalovirus enteritis (Infections and infestations) | 0 | 1
Cytomegalovirus gastroenteritis (Infections and infestations) | 0 | 3
Cytomegalovirus gastrointestinal infection (Infections and infestations) | 0 | 1
Cytomegalovirus hepatitis (Infections and infestations) | 0 | 2
Cytomegalovirus infection (Infections and infestations) | 6 | 48
Dengue fever (Infections and infestations) | 1 | 0
Dermatophytosis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 3
Device related sepsis (Infections and infestations) | 1 | 0
Diabetic foot infection (Infections and infestations) | 1 | 2
Diarrhoea infectious (Infections and infestations) | 1 | 0
Disseminated tuberculosis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 3 | 3
Ear infection (Infections and infestations) | 1 | 0
Encephalitis (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 1
Enteritis infectious (Infections and infestations) | 1 | 0
Enterococcal infection (Infections and infestations) | 1 | 1
Enterococcal sepsis (Infections and infestations) | 1 | 0
Enterocolitis viral (Infections and infestations) | 1 | 0
Epididymitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 3 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 2
Escherichia infection (Infections and infestations) | 1 | 1
Escherichia pyelonephritis (Infections and infestations) | 1 | 1
Escherichia sepsis (Infections and infestations) | 5 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 7
Febrile infection (Infections and infestations) | 1 | 1
Fungal infection (Infections and infestations) | 1 | 1
Fungal sepsis (Infections and infestations) | 0 | 2
Gangrene (Infections and infestations) | 1 | 2
Gastroenteritis (Infections and infestations) | 18 | 23
Gastroenteritis clostridial (Infections and infestations) | 0 | 1
Gastroenteritis cryptosporidial (Infections and infestations) | 0 | 1
Gastroenteritis norovirus (Infections and infestations) | 0 | 6
Gastroenteritis viral (Infections and infestations) | 1 | 3
Gastrointestinal infection (Infections and infestations) | 2 | 1
Groin abscess (Infections and infestations) | 3 | 2
HIV infection (Infections and infestations) | 0 | 1
Haematoma infection (Infections and infestations) | 2 | 0
Hepatic cyst infection (Infections and infestations) | 1 | 0
Hepatitis C (Infections and infestations) | 0 | 1
Hepatitis E (Infections and infestations) | 0 | 1
Hepatitis viral (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 1 | 1
Herpes simplex pneumonia (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 5 | 4
Herpes zoster disseminated (Infections and infestations) | 0 | 1
Ileal gangrene (Infections and infestations) | 0 | 1
Infected lymphocele (Infections and infestations) | 4 | 1
Infected seroma (Infections and infestations) | 1 | 1
Infected skin ulcer (Infections and infestations) | 3 | 2
Infection (Infections and infestations) | 2 | 1
Infectious colitis (Infections and infestations) | 0 | 1
Infectious pleural effusion (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 6 | 5
Intervertebral discitis (Infections and infestations) | 0 | 2
Intestinal sepsis (Infections and infestations) | 1 | 0
Kidney infection (Infections and infestations) | 1 | 2
Klebsiella bacteraemia (Infections and infestations) | 0 | 1
Klebsiella sepsis (Infections and infestations) | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 3
Lung infection (Infections and infestations) | 1 | 2
Medical device site cellulitis (Infections and infestations) | 1 | 0
Medical device site infection (Infections and infestations) | 0 | 1
Meningitis bacterial (Infections and infestations) | 1 | 0
Meningitis cryptococcal (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 1
Nocardiosis (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 2
Oral herpes (Infections and infestations) | 1 | 1
Orchitis (Infections and infestations) | 1 | 3
Osteomyelitis (Infections and infestations) | 5 | 2
Osteomyelitis chronic (Infections and infestations) | 2 | 0
Parvovirus B19 infection (Infections and infestations) | 1 | 0
Perinephric abscess (Infections and infestations) | 2 | 0
Peritonitis (Infections and infestations) | 1 | 0
Peritonsillar abscess (Infections and infestations) | 1 | 1
Pharyngotonsillitis (Infections and infestations) | 0 | 1
Pneumococcal sepsis (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 6 | 3
Pneumonia (Infections and infestations) | 55 | 36
Pneumonia bacterial (Infections and infestations) | 1 | 1
Pneumonia cryptococcal (Infections and infestations) | 0 | 2
Pneumonia cytomegaloviral (Infections and infestations) | 1 | 4
Pneumonia fungal (Infections and infestations) | 0 | 1
Pneumonia haemophilus (Infections and infestations) | 0 | 1
Pneumonia influenzal (Infections and infestations) | 1 | 0
Pneumonia legionella (Infections and infestations) | 1 | 1
Polyomavirus-associated nephropathy (Infections and infestations) | 4 | 10
Postoperative abscess (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 3 | 3
Pseudomembranous colitis (Infections and infestations) | 0 | 1
Pseudomonal bacteraemia (Infections and infestations) | 0 | 1
Pseudomonal sepsis (Infections and infestations) | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 2 | 1
Pyelonephritis (Infections and infestations) | 24 | 33
Pyelonephritis acute (Infections and infestations) | 6 | 13
Pyelonephritis chronic (Infections and infestations) | 1 | 1
Pyuria (Infections and infestations) | 0 | 1
Renal cyst infection (Infections and infestations) | 1 | 3
Renal graft infection (Infections and infestations) | 2 | 0
Respiratory tract infection (Infections and infestations) | 5 | 5
Respiratory tract infection fungal (Infections and infestations) | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0
Rhinovirus infection (Infections and infestations) | 0 | 1
Salmonellosis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 20 | 7
Septic shock (Infections and infestations) | 6 | 8
Sinusitis (Infections and infestations) | 1 | 1
Sinusitis fungal (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 1
Streptococcal sepsis (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 2 | 0
Systemic candida (Infections and infestations) | 0 | 1
Tonsillitis bacterial (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 1 | 1
Transplant abscess (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 0
Tuberculosis gastrointestinal (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 5 | 4
Urinary tract infection (Infections and infestations) | 78 | 93
Urinary tract infection bacterial (Infections and infestations) | 4 | 1
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0
Urinary tract infection fungal (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 23 | 23
Varicella (Infections and infestations) | 0 | 1
Viral diarrhoea (Infections and infestations) | 1 | 1
Viral infection (Infections and infestations) | 2 | 2
Viral myocarditis (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1
Wound abscess (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 5 | 4
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 0
Anaesthetic complication (Injury, poisoning and procedural complications) | 1 | 0
Anastomotic haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Aponeurosis contusion (Injury, poisoning and procedural complications) | 0 | 3
Arterial injury (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 1 | 3
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 | 4
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 2 | 1
Avulsion fracture (Injury, poisoning and procedural complications) | 1 | 0
Complications of transplant surgery (Injury, poisoning and procedural complications) | 1 | 1
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 34 | 28
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Coronary bypass stenosis (Injury, poisoning and procedural complications) | 0 | 1
Delayed graft function (Injury, poisoning and procedural complications) | 7 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 1
Femur fracture (Injury, poisoning and procedural complications) | 2 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1
Graft complication (Injury, poisoning and procedural complications) | 2 | 3
Graft haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Graft loss (Injury, poisoning and procedural complications) | 16 | 12
Graft thrombosis (Injury, poisoning and procedural complications) | 2 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1
Incision site complication (Injury, poisoning and procedural complications) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 8 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Musculoskeletal injury (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 3
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Peripheral arterial reocclusion (Injury, poisoning and procedural complications) | 0 | 1
Perirenal haematoma (Injury, poisoning and procedural complications) | 1 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 3 | 1
Post procedural discharge (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 3 | 1
Post procedural haematuria (Injury, poisoning and procedural complications) | 2 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 4 | 4
Post procedural persistent drain fluid (Injury, poisoning and procedural complications) | 1 | 1
Post procedural urine leak (Injury, poisoning and procedural complications) | 0 | 1
Postoperative fever (Injury, poisoning and procedural complications) | 1 | 0
Postoperative hernia (Injury, poisoning and procedural complications) | 2 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 2
Renal lymphocele (Injury, poisoning and procedural complications) | 3 | 1
Renal transplant torsion (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 1
Scar (Injury, poisoning and procedural complications) | 1 | 0
Scrotal haematoma (Injury, poisoning and procedural complications) | 0 | 2
Seroma (Injury, poisoning and procedural complications) | 5 | 2
Shunt aneurysm (Injury, poisoning and procedural complications) | 2 | 1
Shunt stenosis (Injury, poisoning and procedural complications) | 2 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Stress fracture (Injury, poisoning and procedural complications) | 1 | 0
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 2 | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 2 | 3
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 2
Toxicity to various agents (Injury, poisoning and procedural complications) | 5 | 4
Transplant dysfunction (Injury, poisoning and procedural complications) | 7 | 7
Transplant failure (Injury, poisoning and procedural complications) | 1 | 1
Transplantation complication (Injury, poisoning and procedural complications) | 5 | 1
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Ureteric anastomosis complication (Injury, poisoning and procedural complications) | 1 | 1
Urinary anastomotic leak (Injury, poisoning and procedural complications) | 1 | 1
Vaccination complication (Injury, poisoning and procedural complications) | 1 | 0
Vascular graft complication (Injury, poisoning and procedural complications) | 1 | 1
Vascular graft stenosis (Injury, poisoning and procedural complications) | 0 | 1
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
Wound decomposition (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 10 | 3
Wound secretion (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Anticoagulation drug level above therapeutic (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1
Biopsy kidney (Investigations) | 1 | 0
Blood creatine increased (Investigations) | 2 | 3
Blood creatinine abnormal (Investigations) | 1 | 2
Blood creatinine increased (Investigations) | 50 | 36
Blood glucose increased (Investigations) | 1 | 0
Blood phosphorus decreased (Investigations) | 0 | 1
Blood urea increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 2 | 0
Catheterisation cardiac (Investigations) | 1 | 0
Ejection fraction abnormal (Investigations) | 0 | 1
Electrocardiogram T wave inversion (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1
Haptoglobin decreased (Investigations) | 1 | 0
Immunosuppressant drug level increased (Investigations) | 1 | 0
Inflammatory marker increased (Investigations) | 1 | 2
Liver function test increased (Investigations) | 1 | 0
Norovirus test positive (Investigations) | 1 | 0
Occult blood positive (Investigations) | 1 | 0
Polyomavirus test positive (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 1
Troponin increased (Investigations) | 0 | 1
Urine output decreased (Investigations) | 3 | 0
Weight decreased (Investigations) | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 0 | 2
Calciphylaxis (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2
Dehydration (Metabolism and nutrition disorders) | 6 | 11
Diabetes mellitus (Metabolism and nutrition disorders) | 9 | 10
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 3 | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 5 | 3
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 11 | 10
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 5
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 4
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 1
Intervertebral disc space narrowing (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 2
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 9 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pubic pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 4
Benign gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Bronchioloalveolar carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Epstein-Barr virus associated lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Leydig cell tumour of the testis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Malignant neoplasm of pleura metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Monoclonal gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Papillary tumour of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 4
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 5
Testicular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ataxia (Nervous system disorders) | 0 | 1
Autoimmune encephalopathy (Nervous system disorders) | 0 | 1
Brain injury (Nervous system disorders) | 1 | 0
Brain stem infarction (Nervous system disorders) | 0 | 1
Central nervous system lesion (Nervous system disorders) | 0 | 1
Cerebellar stroke (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Coma (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 3
Encephalopathy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 7
Hyponatraemic seizure (Nervous system disorders) | 1 | 0
Hypotonia (Nervous system disorders) | 1 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 0 | 1
Myelitis transverse (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Neurotoxicity (Nervous system disorders) | 1 | 2
Presyncope (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 3
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Transverse sinus thrombosis (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 2 | 1
Visual field defect (Nervous system disorders) | 1 | 0
Cephalhaematoma (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Device dislocation (Product Issues) | 2 | 1
Device leakage (Product Issues) | 0 | 1
Device malfunction (Product Issues) | 0 | 1
Acute psychosis (Psychiatric disorders) | 1 | 0
Aggression (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Hallucination, visual (Psychiatric disorders) | 0 | 1
Mental disorder (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 2
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 46 | 37
Anuria (Renal and urinary disorders) | 1 | 1
Bladder neck obstruction (Renal and urinary disorders) | 1 | 0
Bladder obstruction (Renal and urinary disorders) | 1 | 0
Bladder perforation (Renal and urinary disorders) | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 2
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0
Diabetic nephropathy (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 5
End stage renal disease (Renal and urinary disorders) | 1 | 0
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 1 | 3
Glomerulonephritis (Renal and urinary disorders) | 1 | 2
Glomerulonephritis chronic (Renal and urinary disorders) | 1 | 0
Glomerulonephritis membranoproliferative (Renal and urinary disorders) | 1 | 1
Glomerulonephritis membranous (Renal and urinary disorders) | 1 | 1
Glycosuria (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 9 | 14
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 9 | 6
Hydroureter (Renal and urinary disorders) | 1 | 0
Hypertonic bladder (Renal and urinary disorders) | 0 | 1
IgM nephropathy (Renal and urinary disorders) | 1 | 0
Ischaemic nephropathy (Renal and urinary disorders) | 0 | 1
Leukocyturia (Renal and urinary disorders) | 0 | 1
Mesangioproliferative glomerulonephritis (Renal and urinary disorders) | 1 | 0
Nephritis (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Nephropathy (Renal and urinary disorders) | 0 | 1
Nephropathy toxic (Renal and urinary disorders) | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1
Obstructive nephropathy (Renal and urinary disorders) | 1 | 1
Oliguria (Renal and urinary disorders) | 2 | 0
Pelvi-ureteric obstruction (Renal and urinary disorders) | 1 | 0
Perinephric collection (Renal and urinary disorders) | 2 | 5
Pollakiuria (Renal and urinary disorders) | 2 | 0
Prerenal failure (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 15 | 3
Pyelocaliectasis (Renal and urinary disorders) | 2 | 1
Renal artery dissection (Renal and urinary disorders) | 1 | 0
Renal artery occlusion (Renal and urinary disorders) | 0 | 1
Renal artery stenosis (Renal and urinary disorders) | 4 | 7
Renal artery thrombosis (Renal and urinary disorders) | 1 | 2
Renal cortical necrosis (Renal and urinary disorders) | 1 | 0
Renal cyst (Renal and urinary disorders) | 0 | 1
Renal cyst haemorrhage (Renal and urinary disorders) | 2 | 1
Renal cyst ruptured (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 3
Renal haematoma (Renal and urinary disorders) | 1 | 1
Renal impairment (Renal and urinary disorders) | 23 | 25
Renal ischaemia (Renal and urinary disorders) | 0 | 1
Renal necrosis (Renal and urinary disorders) | 0 | 1
Renal tubular atrophy (Renal and urinary disorders) | 1 | 1
Renal tubular necrosis (Renal and urinary disorders) | 3 | 5
Renal vein thrombosis (Renal and urinary disorders) | 2 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 1
Ureteric dilatation (Renal and urinary disorders) | 1 | 1
Ureteric obstruction (Renal and urinary disorders) | 3 | 1
Ureteric stenosis (Renal and urinary disorders) | 3 | 6
Urethral obstruction (Renal and urinary disorders) | 1 | 1
Urethral stenosis (Renal and urinary disorders) | 2 | 1
Urge incontinence (Renal and urinary disorders) | 0 | 1
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 | 0
Urinary bladder polyp (Renal and urinary disorders) | 0 | 1
Urinary fistula (Renal and urinary disorders) | 3 | 2
Urinary incontinence (Renal and urinary disorders) | 9 | 1
Urinary retention (Renal and urinary disorders) | 1 | 8
Urinary tract obstruction (Renal and urinary disorders) | 2 | 4
Urinoma (Renal and urinary disorders) | 1 | 0
Vesicoureteric reflux (Renal and urinary disorders) | 1 | 0
Acquired hydrocele (Reproductive system and breast disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 3
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 3 | 4
Scrotal oedema (Reproductive system and breast disorders) | 1 | 0
Testicular oedema (Reproductive system and breast disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 7
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 17 | 6
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Capillaritis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Neuropathic ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Peau d'orange (Skin and subcutaneous tissue disorders) | 1 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin oedema (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1
Loss of personal independence in daily activities (Social circumstances) | 1 | 0
Walking disability (Social circumstances) | 1 | 0
Arteriovenous fistula operation (Surgical and medical procedures) | 0 | 1
Orchidectomy (Surgical and medical procedures) | 1 | 0
Accelerated hypertension (Vascular disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0
Aortic perforation (Vascular disorders) | 0 | 1
Arterial stenosis (Vascular disorders) | 1 | 0
Arterial thrombosis (Vascular disorders) | 1 | 0
Arteriovenous fistula (Vascular disorders) | 1 | 1
Artery dissection (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 20 | 12
Embolism venous (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 3
Hypertension (Vascular disorders) | 2 | 6
Hypertensive crisis (Vascular disorders) | 3 | 5
Hypertensive emergency (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 3 | 8
Intermittent claudication (Vascular disorders) | 0 | 1
Lymphocele (Vascular disorders) | 34 | 21
Lymphorrhoea (Vascular disorders) | 3 | 0
Malignant hypertension (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1
Pelvic venous thrombosis (Vascular disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 1
Peripheral artery stenosis (Vascular disorders) | 0 | 2
Peripheral artery thrombosis (Vascular disorders) | 2 | 1
Peripheral ischaemia (Vascular disorders) | 2 | 1
Phlebitis (Vascular disorders) | 1 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 2
Thrombophlebitis superficial (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 2 | 0
Varicose ulceration (Vascular disorders) | 1 | 0
Venous stenosis (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 1 | 3
Venous thrombosis limb (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus Plus@Reduced CNI (N=1014) | MPA Plus Standard@CNI (N=1012)
Anaemia (Blood and lymphatic system disorders) | 227 | 238
Leukocytosis (Blood and lymphatic system disorders) | 24 | 58
Leukopenia (Blood and lymphatic system disorders) | 94 | 194
Polycythaemia (Blood and lymphatic system disorders) | 52 | 42
Thrombocytopenia (Blood and lymphatic system disorders) | 74 | 41
Tachycardia (Cardiac disorders) | 53 | 52
Abdominal pain (Gastrointestinal disorders) | 94 | 104
Abdominal pain upper (Gastrointestinal disorders) | 39 | 62
Constipation (Gastrointestinal disorders) | 245 | 242
Diarrhoea (Gastrointestinal disorders) | 242 | 318
Nausea (Gastrointestinal disorders) | 191 | 225
Vomiting (Gastrointestinal disorders) | 120 | 140
Fatigue (General disorders) | 59 | 64
Oedema peripheral (General disorders) | 347 | 244
Pyrexia (General disorders) | 112 | 132
BK virus infection (Infections and infestations) | 56 | 101
Cytomegalovirus infection (Infections and infestations) | 24 | 93
Nasopharyngitis (Infections and infestations) | 110 | 117
Upper respiratory tract infection (Infections and infestations) | 81 | 102
Urinary tract infection (Infections and infestations) | 219 | 249
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 63 | 54
Incision site pain (Injury, poisoning and procedural complications) | 51 | 61
Procedural pain (Injury, poisoning and procedural complications) | 90 | 99
Blood creatinine increased (Investigations) | 141 | 133
Weight increased (Investigations) | 38 | 66
Diabetes mellitus (Metabolism and nutrition disorders) | 133 | 120
Dyslipidaemia (Metabolism and nutrition disorders) | 98 | 57
Hypercalcaemia (Metabolism and nutrition disorders) | 39 | 67
Hypercholesterolaemia (Metabolism and nutrition disorders) | 103 | 61
Hyperglycaemia (Metabolism and nutrition disorders) | 140 | 144
Hyperkalaemia (Metabolism and nutrition disorders) | 164 | 184
Hyperlipidaemia (Metabolism and nutrition disorders) | 135 | 75
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 58 | 24
Hyperuricaemia (Metabolism and nutrition disorders) | 49 | 64
Hypocalcaemia (Metabolism and nutrition disorders) | 109 | 98
Hypokalaemia (Metabolism and nutrition disorders) | 148 | 87
Hypomagnesaemia (Metabolism and nutrition disorders) | 134 | 168
Hypophosphataemia (Metabolism and nutrition disorders) | 190 | 167
Metabolic acidosis (Metabolism and nutrition disorders) | 77 | 98
Vitamin D deficiency (Metabolism and nutrition disorders) | 53 | 57
Arthralgia (Musculoskeletal and connective tissue disorders) | 63 | 65
Back pain (Musculoskeletal and connective tissue disorders) | 93 | 98
Pain in extremity (Musculoskeletal and connective tissue disorders) | 66 | 61
Dizziness (Nervous system disorders) | 51 | 54
Headache (Nervous system disorders) | 133 | 113
Tremor (Nervous system disorders) | 100 | 145
Anxiety (Psychiatric disorders) | 51 | 59
Insomnia (Psychiatric disorders) | 100 | 138
Dysuria (Renal and urinary disorders) | 60 | 74
Haematuria (Renal and urinary disorders) | 102 | 101
Proteinuria (Renal and urinary disorders) | 131 | 69
Cough (Respiratory, thoracic and mediastinal disorders) | 86 | 102
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 73 | 70
Acne (Skin and subcutaneous tissue disorders) | 56 | 37
Alopecia (Skin and subcutaneous tissue disorders) | 27 | 59
Hypertension (Vascular disorders) | 240 | 230
Hypotension (Vascular disorders) | 62 | 78

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-07-14): https://cdn.clinicaltrials.gov/large-docs/19/NCT01950819/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-27): https://cdn.clinicaltrials.gov/large-docs/19/NCT01950819/SAP_001.pdf